CLINICAL TRIAL: NCT00085059
Title: Early Phase II Study On BNCT In Metastatic Malignant Melanoma Using The Boron Carrier BPA
Brief Title: Boron Neutron Capture Therapy Using Boronophenylalanine-Fructose Complex in Treating Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-11011; EORTC-11011
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — 4-boronophenylalanine-fructose

INTERVENTIONS:
Drug: boronophenylalanine-fructose complex

SUMMARY:
RATIONALE: Boron neutron capture therapy using boronophenylalanine-fructose complex may kill tumor cells without harming normal tissue.

PURPOSE: This phase II trial is studying how well boron neutron capture therapy using boronophenylalanine-fructose complex works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the therapeutic activity and efficacy of boron neutron capture therapy using boronophenylalanine-fructose complex in patients with metastatic melanoma.
* Determine the objective local response in patients treated with this regimen.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the duration of local response and time to local progression in patients treated with this regimen.
* Determine the dose-response relationship at the per-lesion level in patients treated with this regimen.
* Determine the safety of this regimen in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive boronophenylalanine-fructose complex IV over 90 minutes followed by boron neutron capture therapy on days 1 and 2.

Patients are followed at 1 and 6 weeks and then every 8 weeks thereafter. In the event of disease progression, patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 16-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Metastatic disease

    * Brain metastases, skin metastases, or soft tissue metastases of the head and neck or the extremities
  * Accessible lesion(s) for boron neutron capture therapy (BNCT)
  * No clear progression of disease at other sites than the ones intended for treatment with surgery and/or BNCT
* Measurable disease by MRI within the past 4 weeks

  * Lesion(s) ≥ 10 mm in diameter
* Indication for palliative radiotherapy that is intended to be delivered as BNCT

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin ≤ 2.5 times upper limit of normal (ULN)*
* Transaminases ≤ 2.5 times ULN*
* Alkaline phosphatase ≤ 2.5 times ULN* NOTE: *Unless due to reversible reaction to antiseizure medication

Renal

* Creatinine ≤ 2.5 times ULN
* Blood urea nitrogen ≤ 2.5 times ULN

Cardiovascular

* No congestive heart failure
* No newly diagnosed or unstable angina pectoris
* No uncontrolled arrhythmias
* No uncontrolled conduction defects
* No recent coronary artery disease
* No other severe heart disease

Pulmonary

* No severe pulmonary disease, including severe obstructive or restrictive lung disease

Other

* No history of phenylketonuria
* No severe gastrointestinal disease
* No active peptic ulcer disease
* No uncontrolled endocrine disease
* No pre-existing serious mental or organic brain disease (e.g., epilepsy)
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* Able to travel to the Netherlands via public transportation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunologic or biologic therapy
* No concurrent colony-stimulating factors (e.g., epoetin alfa or filgrastim [G-CSF])

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No prior radiotherapy to site(s) proposed for study treatment
* No other concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* Recovered from all prior anti-tumor therapy (excluding alopecia and sensitive peripheral neuropathy ≤ grade 2)
* No other concurrent anticancer therapy
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Best response to treatment as measured by RECIST every 8 weeks at completion of study treatment

SECONDARY OUTCOMES:
Overall survival as measured every 8 weeks at completion of study treatment
Duration of local response as measured by Kaplan Meier every 8 weeks after completion of study treatment
Time to local progression measured every 8 weeks after completion of study treatment
Acute toxicity as measured by Common Toxicity Criteria AE v 3.0 1- 6 weeks after completion of treatment
Late toxicity as measured by RTOG and EORTC week 6 and thereafter upon completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wittig, Study Chair — Universitaetsklinikum Essen
Locations (1):
- Universitaetsklinikum Essen, Essen, Germany

REFERENCES:
- [Background] Wittig A, Moss RL, Stecher-Rasmussen F, Appelman K, Rassow J, Roca A, Sauerwein W. Neutron activation of patients following boron neutron capture therapy of brain tumors at the high flux reactor (HFR) Petten (EORTC Trials 11961 and 11011). Strahlenther Onkol. 2005 Dec;181(12):774-82. doi: 10.1007/s00066-005-1433-4. PMID 16362787